CLINICAL TRIAL: NCT00076726
Title: A Randomized, Double-Masked, Placebo-Controlled, Multicenter Study of the Safety and Efficacy of Infliximab in Subjects With Giant Cell Arteritis
Brief Title: A Study of the Safety and Effectiveness of Infliximab (Remicade) in Patients With Giant Cell Arteritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis, infliximab did not reduce number of first relapses in GCA or cumulative glucocorticosteroid dosage
Sponsor: Centocor, Inc. (Industry)
Collaborators: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003139
Record Dates: First submitted 2004-02-02; First posted 2004-02-04 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Giant Cell Arteritis
Keywords: Giant Cell Arteritis; infliximab
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Infliximab

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy (effectiveness) of Infliximab (Remicade) in patients with Giant Cell Arteritis. Infliximab (Remicade) targets specific proteins in the body's immune system to help control the development of inflammation to help reduce painful disease.

DETAILED DESCRIPTION:
The purpose of this study is to see if infliximab is safe and effective in treating GCA. Currently, the only treatment for GCA is prednisone. GCA is a long lasting inflammatory disease. The cause is unknown. It may affect all the arteries, but it focuses on the big vessels such as those around the heart, the vessels in the neck and head, and their major branches. It can lead to vision loss, blindness, stroke, stenosis (narrowing of blood vessels) and aneurysms (a weakening in the lining of the blood vessel wall, which may eventually lead to rupture of the blood vessel). The damage to the arteries is caused by an immune response. A naturally occurring substance in the immune system called "tumor necrosis factor alpha" (TNFa) plays a significant role in this immune response against the blood vessels. This response is thought to cause the long-lasting inflammation (irritation and swelling of the vessels). By blocking the effect of TNFa we think that we may reduce the signs and symptoms associated with GCA. This trial will study patients who are stable on prednisone treatment by evaluating whether infliximab can control their symptoms as the dose of prednisone is reduced. Patients will receive infusions of either 5mg/kg of infliximab or placebo at weeks 0, 2, 6, 14, 22, 30, 38, and 46. Safety evaluations will be performed at specified intervals throughout the study and will consist of laboratory tests, vital signs (such as blood pressure), physical examinations and the occurrence and severity of adverse events as well as other study specific procedures. Patients will receive receive infusions of either 5mg/kg infliximab or placebo infusions at weeks 0, 2, 6, 14, 22, 30, 38, and 46.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a diagnosis of Giant Cell Arteritis (GCA)
* Patients who have a diagnosis of GCA of = 4 weeks' duration
* Patients who are receiving = 40 mg/day of prednisone/prednisolone Exclusion Criteria:
* Patients must not have a prior diagnosis of GCA > 4 weeks
* Patients must not have failed to respond to glucocorticosteroid therapy within 5 days of initiation of therapy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-11; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
The proportion of relapse-free patients through Week 22 .

SECONDARY OUTCOMES:
Proportion of relapse-free subjects through Week 54, time to first relapse, levels of biochemical markers of inflammation and disease activity (eg, ESR, C-reactive protein [CRP], interleukin [IL]-6) , cumulative dose of prednisone (or equivalents)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Hoffman GS, Cid MC, Rendt-Zagar KE, Merkel PA, Weyand CM, Stone JH, Salvarani C, Xu W, Visvanathan S, Rahman MU; Infliximab-GCA Study Group. Infliximab for maintenance of glucocorticosteroid-induced remission of giant cell arteritis: a randomized trial. Ann Intern Med. 2007 May 1;146(9):621-30. doi: 10.7326/0003-4819-146-9-200705010-00004. PMID 17470830
- [Derived] Visvanathan S, Rahman MU, Hoffman GS, Xu S, Garcia-Martinez A, Segarra M, Lozano E, Espigol-Frigole G, Hernandez-Rodriguez J, Cid MC. Tissue and serum markers of inflammation during the follow-up of patients with giant-cell arteritis--a prospective longitudinal study. Rheumatology (Oxford). 2011 Nov;50(11):2061-70. doi: 10.1093/rheumatology/ker163. Epub 2011 Aug 25. PMID 21873264
- See also: A Randomized, Double-masked, Placebo-controlled, Multicenter Study of the Safety and Efficacy of Infliximab in Subjects with Giant Cell Arteritis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=145&filename=CR003139_CSR.pdf